CLINICAL TRIAL: NCT02926170
Title: Rivaroxaban Versus Acenocumarol for Secondary Thromboprophylaxis in Patients With Antiphospholipid Syndrome: a Randomized, Prospective, Phase III Study. Analysis of Stratification Prognostic Factors
Brief Title: Rivaroxaban for Patients With Antiphospholipid Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-019764-36
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Rivaroxaban; Acenocoumarol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rivaroxaban (Experimental): Rivaroxaban 20 mg per day
  Interventions: Drug: Rivaroxaban
- acenocumarol (Active Comparator): INR adjusted dose
  Interventions: Drug: acenocumarol

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban will be started at 20 mg/day. Dose will be adjusted according to Cr Clearance. Cr Clearance 30-49 ml/min will receive 15 mg/day.
  Other Names: XARELTO
  Arms: rivaroxaban
Drug: acenocumarol — Doses will be adjusted according to INR
  Other Names: SINTROM
  Arms: acenocumarol

SUMMARY:
Long-term anticoagulation is widely used for secondary thromboprophylaxis in the antiphospholipid syndrome (APS) due to the high risk of recurrent events. Currently anticoagulation with vitamin K antagonists (VKAs) is the standard of care but have unpredictable pharmacodynamic properties that requiere monitoring for dose adjustment. Rivaroxaban, an orally active direct factor Xa inhibitor, has been shown to be effective and safe compared with warfarin for the treatment of venous thromboembolism and non valvular atrial fibrillation in major RCTs. No studies had been published in APS.The aim of the study is to investigate the efficacy and safety of rivaroxaban in preventing recurrent thrombosis in patients with APS compared with acenocoumarol

DETAILED DESCRIPTION:
This is a phase 3 randomized, multicenter, non-inferiority open-label RCT. 190 eligible APS patients with arterial or venous thrombotic history receiving acenocoumarol will be stratified according the presence of SLE and venous/arterial thrombotic history and randomized (1:1) either to continue vitamin K antagonists (standard of care, normalized ratio (INR) 2-3 or 2.5 to 3.5 in those with recurrent thrombotic episodes) or to switch to rivaroxaban (20 mg/day). The primary efficacy outcome is the development of any thrombotic event during the study period. Secondary efficacy outcomes include time to thrombosis, type of thrombosis (arterial or venous), overall causes of death, evaluation of a prognostic biomarker panel of recurrent thrombosis. The primary safety outcome will be major bleeding. Secondary safety outcomes include any adverse event and minor bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thrombotic antiphsopholipd syndrome
* Treated with acenocumarol for a minimum period of 6 months
* Positivity for Lupus anticoagulant and/or anti-cardiolipin or anti-B2GPI antibodies IgG or IgM≥40

Exclusion Criteria:

* Major haemorrhage (cerebral or gastrointestinal) within the previous 6 months
* Neurosurgery within the previous 4 weeks
* Any surgery within the previous 10 days
* Active peptic ulcus
* ALT or GPT >120 UI/mL non-lupus related in the previous 30 days
* Platelets <30x10E9 in the previous 30 days
* Recent diagnosed malignancy
* Any criteria listed in the summary of the produt characterisitcs (SPC)
* Renal disease with a creatinine clearance <30 mL/min or with a known uncontrolled renal disease
* Concomitant administration of drugs that could interfere with CYP3A4

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Developement of a new thrombotic event (arterial or venous), confirmed by appropiate imaging studies | 36 months
  Stroke or transient ischemic attack, myocardial infarction, peripheral arterial thrombosis, cerebral vein thrombosis, deep-vein thrombosis, or pulmonary embolism) that was confirmed by adjudication
Incidence of major bleeding | 36 months
  Major bleeding is defined as clinically overt bleeding associated with any of the following: fatal bleeding causing death, involvement of a critical anatomic site (intracranial, spinal, intraocular, pericardial, articular, retroperitoneal, or intramuscular with compartment syndrome) or need for surgery or angiographic intervention to stop haemorrhage, fall in haemoglobin concentration of at least 20 g/L in 24 hours, and/or requiring non-planned transfusion of ≥2 units of packed red blood cells or whole blood

SECONDARY OUTCOMES:
Incidence of any treatment-Emergent Adverse events | 36 months
  i) all adverse events; ii) serious adverse events (SAE); iii) all bleeding events; iv) overall causes of death
Death due to thrombotic events | 36 months
  Death as result of a thrombotic event
Time to the first thrombotic event | 36 months
  Time (months) from the treatment onset up to the thrombotic event
Location of thrombotic events | 36 months
  Location (arterial or venous) whenre the thrombotic event occurred
Evaluation of a prognostic biomarker panel | 36 months
  Measuremnt of D-dimer, P-selectine and Von-willebrand factor

CONTACTS AND LOCATIONS:
Overall Officials: Josefina Cortes, MD,pHD, Principal Investigator — Vall d'Hebron Research Institute
Locations (1):
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided